CLINICAL TRIAL: NCT04149665
Title: Compliance of Recommended Semirecumbent Position in Ventilated Patients
Brief Title: Semirecumbent Position by Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bürgerspital Solothurn (Other)
Responsible Party: Principal Investigator, Marcos Delgado, Principal investigator, Bürgerspital Solothurn
Other Study IDs: Req-2019-01052
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Mechanical Ventilation Complication; Ventilator Associated Pneumonia; Compliance, Treatment
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: simple blind observation — Device that measures continuously the angle of bed by mechanical Ventilation to assess the time the bed is above 35°.

SUMMARY:
It's based in an observational trial in mechanical ventilated patients. The investigators assess the head of bed elevation angle in the routine treatment of the unit. The investigators decide to assess the time the patient has a semirecumbent position >35°.

DETAILED DESCRIPTION:
A Semirecumbent-bed position in mechanical ventilated patients is recommended in every international guidelines in order to avoiding Ventilator Associated Pneumonia (VAP). Despite being a simple and cheap measure, the literature describe a low compliance. Globally, every intensive care unit tends to use different maneuvers that help or improve compliance of this recommendation. However, there are multiple factors in daily work that hinder compliance. Before taking actions, it would be convenient to know the current state of the unit.

Investigators aim to evaluate the quality with which the recommendation is carried out in the unit in order to maintain a semirecumbent position. To conduct the Trial it will be used a device that measures continuously (every 5 minutes) the angle of the bed without giving any information to caregivers. Once patients are extubated the data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Every ventilated patients

Exclusion Criteria:

* Patients excluded are those lower that 18 years old or neurocritical patients that require flat position.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to include every mechanical ventilated patients any reason.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-01-11 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Compliance of semirecumbent position in mechanical ventilated patients | November 2019 to April 2020
  Assess how long are mechanical ventilated patient with a head of bed elevation above 35°.

SECONDARY OUTCOMES:
Demographic and disease characteristics of involved patients. | November 2019 to April 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Bürgerspital Solothurn, Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kollef MH. Ventilator-associated pneumonia. A multivariate analysis. JAMA. 1993 Oct 27;270(16):1965-70. PMID 8411554
- [Background] Deye N, Lellouche F, Maggiore SM, Taille S, Demoule A, L'Her E, Galia F, Harf A, Mancebo J, Brochard L. The semi-seated position slightly reduces the effort to breathe during difficult weaning. Intensive Care Med. 2013 Jan;39(1):85-92. doi: 10.1007/s00134-012-2727-5. Epub 2012 Oct 24. PMID 23093247
- [Background] Drakulovic MB, Torres A, Bauer TT, Nicolas JM, Nogue S, Ferrer M. Supine body position as a risk factor for nosocomial pneumonia in mechanically ventilated patients: a randomised trial. Lancet. 1999 Nov 27;354(9193):1851-8. doi: 10.1016/S0140-6736(98)12251-1. PMID 10584721
- [Background] van Nieuwenhoven CA, Vandenbroucke-Grauls C, van Tiel FH, Joore HC, van Schijndel RJ, van der Tweel I, Ramsay G, Bonten MJ. Feasibility and effects of the semirecumbent position to prevent ventilator-associated pneumonia: a randomized study. Crit Care Med. 2006 Feb;34(2):396-402. doi: 10.1097/01.ccm.0000198529.76602.5e. PMID 16424720
- [Background] Alexiou VG, Ierodiakonou V, Dimopoulos G, Falagas ME. Impact of patient position on the incidence of ventilator-associated pneumonia: a meta-analysis of randomized controlled trials. J Crit Care. 2009 Dec;24(4):515-22. doi: 10.1016/j.jcrc.2008.09.003. Epub 2009 Feb 13. PMID 19327314
- [Result] Vincent JL, Bihari DJ, Suter PM, Bruining HA, White J, Nicolas-Chanoin MH, Wolff M, Spencer RC, Hemmer M. The prevalence of nosocomial infection in intensive care units in Europe. Results of the European Prevalence of Infection in Intensive Care (EPIC) Study. EPIC International Advisory Committee. JAMA. 1995 Aug 23-30;274(8):639-44. PMID 7637145